CLINICAL TRIAL: NCT00672087
Title: Diagnostic Challenges in IC (and Male CPPS)
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Jordan Dimitrakoff, MD, PhD, Director of Urogynecology and Chronic Pelvic Pain Lab, Beth Israel Deaconess Medical Center and Harvard Medical School, Boston, MA
Other Study IDs: 2010P000229; R01DK065990 (NIH)
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2014-02

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome; Chronic Bacterial Prostatitis; Asymptomatic Inflammatory Prostatitis; Painful Bladder Syndrome; Cystitis, Interstitial
Keywords: Chronic Prostatitis with Chronic Pelvic Pain Syndrome; Chronic Bacterial Prostatitis; Asymptomatic Inflammatory Prostatitis; Painful Bladder Syndrome; Cystitis, Interstitial
MeSH Terms: conditions — Prostatitis; Cystitis, Interstitial | interventions — Genome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, whole blood, serum, white cells, urine, prostatic fluid, prostate/bladder tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: Chronic prostatitis/chronic pelvic pain syndrome patients
  Interventions: Genetic: Genomic and proteomic biomarker discovery
- B: Painful bladder syndrome/interstitial cystitis patients
  Interventions: Genetic: Genomic and proteomic biomarker discovery
- C: Asymptomatic controls
  Interventions: Genetic: Genomic and proteomic biomarker discovery

INTERVENTIONS:
Genetic: Genomic and proteomic biomarker discovery — Discovery of novel biomarkers for CP/CPPS and PBS/IC using genomic and proteomic methods

SUMMARY:
The etiology and pathogenesis of interstitial cystitis (IC) and its related condition in men, chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) has remained elusive. This has hampered development of mechanistic treatment strategies for these common, chronic and distressing medical conditions. We believe that IC and perhaps CP/CPPS are a spectrum of complex but inter-related genetic and acquired diseases resulting from the interaction of several genes regulating immune/inflammatory and neurogenic parameters and environmental factors/circumstances or exposure, culminating in the combination of pain, frequency, urgency and sexual specific symptoms. New research has delineated the dynamic and powerful association of the immune and neurogenic system in pain activation. An immune-modulated neurogenic model of IC illuminating the action of immune derived substances and pain related substances might be important in discovering the determinants of pain, voiding dysfunction and gender specific sexual problems. This inter-related dynamic model of IC disease pathogenesis could be explored for potential avenues leading to novel diagnostic and treatment strategies. We plan to identify and evaluate the sensitivity and specificity of several novel nerve and inflammation related markers in the diagnosis and follow up of IC (and CP/CPPS). By correlating the levels of urine immune and pain related substances to disease mechanisms, severity and progression, we may be able to create a human disease specific model for diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant has signed and dated the appropriate Informed Consent document.
* Participant must have had symptoms of discomfort or pain in the pelvic region for at least a three (3) month period within the last six (6) months.

Exclusion Criteria:

* Major structural/anatomical urinary tract abnormalities
* Underlying inborn conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary university medical centers and primary care clinic
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2003-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan D Dimitrakoff, MD, PhD, Study Chair — Harvard Medical School, Boston, MA
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Dimitrakov J, Kroenke K, Steers WD, Berde C, Zurakowski D, Freeman MR, Jackson JL. Pharmacologic management of painful bladder syndrome/interstitial cystitis: a systematic review. Arch Intern Med. 2007 Oct 8;167(18):1922-9. doi: 10.1001/archinte.167.18.1922. PMID 17923590
- [Background] Dimitrakov JD, Kaplan SA, Kroenke K, Jackson JL, Freeman MR. Management of chronic prostatitis/chronic pelvic pain syndrome: an evidence-based approach. Urology. 2006 May;67(5):881-8. doi: 10.1016/j.urology.2005.12.015. No abstract available. PMID 16698346
- [Background] Allsop SA, Erstad DJ, Brook K, Bhai SF, Cohen JM, Dimitrakoff JD. The DABBEC phenotyping system: towards a mechanistic understanding of CP/CPPS. Nat Rev Urol. 2011 Feb;8(2):107-13. doi: 10.1038/nrurol.2010.227. Epub 2011 Jan 18. PMID 21243018
- [Background] Strauss AC, Dimitrakov JD. New treatments for chronic prostatitis/chronic pelvic pain syndrome. Nat Rev Urol. 2010 Mar;7(3):127-35. doi: 10.1038/nrurol.2010.4. Epub 2010 Feb 9. PMID 20142810
- [Result] Dimitrakov J, Joffe HV, Soldin SJ, Bolus R, Buffington CA, Nickel JC. Adrenocortical hormone abnormalities in men with chronic prostatitis/chronic pelvic pain syndrome. Urology. 2008 Feb;71(2):261-6. doi: 10.1016/j.urology.2007.09.025. PMID 18308097